CLINICAL TRIAL: NCT02763956
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Efficacy Study of the Gelstix™ Device to Treat Chronic Discogenic Low Back Pain
Brief Title: RCT Study of the Gelstix™ Device to Treat Chronic Discogenic Low Back Pain GelStix Study
Acronym: GelStix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Regionale di Lugano (Other)
Collaborators: Rijnstate Ziekenhuis, Arnhem, The Netherlands (Unknown); Paolo Maino, Sponsor-Investigator (Unknown)
Responsible Party: Principal Investigator, Eva Koetsier MD PhD LLM, MD PhD LLM, Ospedale Regionale di Lugano
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GelStix-SW/ NSI-TD-003
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
Keywords: Gelstix, Hydrogel
MeSH Terms: interventions — Bandages, Hydrocolloid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gelstix (Experimental): The intradiscal insertion of the GelStix™ Nucleus Augmentation Device.
  Interventions: Device: GelStix™ Nucleus Augmentation Device
- Placebo (Placebo Comparator): Intradiscal saline solution (1 mL NaCl 0.9%) injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: GelStix™ Nucleus Augmentation Device — Intradiscal Gelstix insertion
  Other Names: Hydrogel
  Arms: Gelstix
Other: Placebo — Intradiscal saline injection
  Other Names: Saline, NaCl 0,9%
  Arms: Placebo

SUMMARY:
Degenerative Disc Disease is one of the most common spinal pathologies, affecting up to 10-15 % of adults. The purpose of this study is to evaluate the efficacy of treatment with the GelStix™ device in a patient population with discogenic pain that had no benefit from conservative care.

DETAILED DESCRIPTION:
Degenerative Disc Disease (DDD) is one of the most common spinal pathologies, affecting up to 10-15 % of adults. The degeneration is associated with diminished water-binding capabilities of the nucleus pulpous leading to disc dehydration, volume reduction, changes in cellular activity, biomechanical changes and painful symptoms. Patients are initially treated with non-surgical pain-management techniques, such as anti-inflammatory medications and physical therapy, but these therapies often provide only temporary relief. When non-surgical intervention fails, fusion or total disc arthroplasty are often prescribed, both of which are highly invasive surgeries with significant associated morbidity. Clearly, a meaningful solution for the treatment gap existing between conservative care and invasive surgical intervention is needed.

The purpose of this study is to evaluate the efficacy of treatment with the GelStix™ device in a patient population that had no benefit from conservative care.

The primary objective of this study is to quantify the reduction in lumbar pain in a GelStix™ treatment group compared with a control group receiving a saline solution injection as placebo.

The secondary objectives are to assess:

* Disability, using the Oswestry Disability Index (ODI)
* Quality of life (QoL), quantified with the European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L).
* The Patient's Global Impression of Change (PGIC) scale. This scale assesses the patient's own evaluation of improvement or deterioration over time on a 7-point Likert Scale rated from 'very much improved' to 'very much worse'.
* The use of pain medication
* The disc degeneration process will be assessed by means of MRI twelve months after treatment compared to baseline. Pfirrmann grade, disc height, and the presence of high intensity zones, Modic signs, and Schmorl's nodes will be recorded.
* The incidence and severity of complications and adverse events

The total expected number of patients to be randomized is 72. Taking into account a relevant difference of 1.5 between groups on the NRS, with an SD of 2, 30 patients per group (60 patients in total) will be required to detect a statistically significant difference with a power of 80% at an alpha of 5% (two-tailed) for unpaired Student's T test. Taking into account a 20% drop out rate, 72 patients are expected to be randomized for this study.

The estimated duration for the investigational plan (from start of screening of first participant to end of follow-up of last participant) is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* discogenic pain caused by one or two levels of degenerative disc disease, confirmed by MRI and positive discography
* failure to have symptoms resolved or reduced following at least 12 weeks of conservative care (pain medication and/or physical therapy)
* negative medial branches block results
* baseline Numeric Rating Scale (NRS) pain score ≥5/10

Exclusion Criteria:

* radiculopathy
* disc herniations
* annular tear (greater than Grade 4 Modified Dallas Grading)
* coagulopathy or oral anticoagulant therapy (except low-dose acetylsalicylic acid) in conditions that do not allow for a temporary discontinuation
* previous lumbar surgery
* disc height less than 5 mm at the treatment level or less than 50% the original height
* BMI (Body Mass Index (kg/m2) of ≥ 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-04; Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Lumbar Pain intensity measured on Numeric Rating Scale | The mean NRS scores on the pain diary will be measured at baseline, and at one week, and one, three, six (primary outcome) and twelve months.
  Pain intensity will be assessed employing an 11-point (i.e. 0-10) NRS with 0 meaning 'no pain' and '10' meaning 'worst possible pain'. Three times daily pain scores will be assessed for five consecutive days around the intended measurement time.

SECONDARY OUTCOMES:
Changes in disability measured by the Owestry Disability Index | The ODI is completed at baseline, and at three, six and twelve months.
  The ODI is a self-administered questionnaire, assessing the patient's level of pain and function during basic activities of daily living such as walking, personal care, standing, sleeping, etc.
Changes in health related quality of life measured by EuroQualityOfLife-5 dimensions questionnaire | The EQ-5D-5L will be completed at baseline and at three, six and twelve months.
  This questionnaire assesses health related quality of life in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.49 Additionally, the EuroQol Visual Analogue Scale (EQ VAS) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine'.
The Patient's Global Impression of Change (PGIC) scale | The Patient's Global Impression of Change (PGIC) scale will be measured at three, six and twelve months.
  This scale assesses the patient's own evaluation of improvement or deterioration over time on a 7-point Likert Scale rated from 'very much improved' to 'very much worse'.
Pain medication | The use of pain medication will be assessed as the intake of analgesics at baseline, at one week, and at one, three, six and twelve months.
  Reliance on medication to relieve pain: type and dose of analgesics
The disc degeneration process | The disc degeneration process will be assessed by means of MRI twelve months after treatment compared to baseline.
  Pfirrmann grade, disc height, and the presence of high intensity zones (HIZ), Modic signs, and Schmorl's nodes will be recorded.
The incidence and severity of complications and adverse events | The incidence and severity of complications and adverse events are assessed at any time point in the study up to one year follow up.
  The safety outcome of this study is the incidence and severity of complications and adverse events (AE's) including procedure-related complications at any time point in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Koetsier, MD PhD LLM, Principal Investigator — Centro Terapia del Dolore, EOC Lugano
Locations (2):
- Rijnstate Ziekenhuis, Arnhem, Netherlands
- EOC Lugano, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Koetsier E, van Kuijk SMJ, Maino P, Dukanac J, Scascighini L, Cianfoni A, Scarone P, Kuhlen DE, Hollman MW, Kallewaard JW. Efficacy of the Gelstix nucleus augmentation device for the treatment of chronic discogenic low back pain: protocol for a randomised, sham-controlled, double-blind, multicentre trial. BMJ Open. 2022 Mar 30;12(3):e053772. doi: 10.1136/bmjopen-2021-053772. PMID 35354635